CLINICAL TRIAL: NCT01413958
Title: A Randomized, Placebo-Controlled Trial to Evaluate the Effects of Phenylephrine HCl 30 mg Extended-Release Tablets on Nasal Congestion in Subjects With Allergic Rhinitis
Brief Title: Effects of Phenylephrine Extended-Release Tablets on Allergy-Related Nasal Congestion (P08498 AM1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18125; CL2011-06 (Other: CHC protocol number); P08498 (Other: Merck)
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Results first posted 2013-01-29 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-02

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Nasal Decongestants; Rhinitis, Allergic, Seasonal; Rhinitis; Nose Conditions; Respiratory Tract Diseases; Phenylephrine
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis; Respiratory Tract Diseases | interventions — Phenylephrine; Loratadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phenylephrine (Experimental)
  Interventions: Drug: Phenylephrine; Drug: Loratadine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Loratadine

INTERVENTIONS:
Drug: Phenylephrine — Phenylephrine hydrochloride 30-mg extended-release tablets, one tablet every 12 hours for 7 days
  Other Names: SCH 002063; MK-9314
  Arms: Phenylephrine
Drug: Placebo — Placebo to phenylephrine hydrochloride 30-mg extended release tablets, one tablet every 12 hours for 7 days
  Arms: Placebo
Drug: Loratadine — Loratadine, 10 mg, once daily as rescue medication, only if needed for intolerable allergic rhinitis symptoms
  Other Names: Claritin®

SUMMARY:
This study will compare the nasal congestion symptom relief of phenylephrine extended release tablets and placebo in participants with allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Understands study procedures and agrees to participate by giving signed consent form
* Male or female, aged 18 years or older, at the Screening Visit.
* Female participants must demonstrate a negative urine pregnancy test, at Screening (Visit 1) and Visit 2 (prior to randomization) and agree to use (and/or have their partner use) 2 acceptable methods of birth control beginning at the Screening visit and throughout the study and until 2 weeks after the last dose of study drug in the last treatment period. Acceptable methods of birth control are abstinence, or two of the following:

  * hormonal contraceptives (with documented use for at least 30 days prior to Screening )
  * intrauterine device (IUD)
  * diaphragm with spermicide
  * contraceptive sponge
  * condom
  * vasectomy
* Willing to stop use of current decongestant and allergy medications during the trial
* Documented or self-reported history of allergic rhinitis caused by fall pollen within the last 4 years

and documented or self-reported symptoms over at least the last 2 fall allergy seasons

* Documented skin testing (prick with wheal ≥3 mm larger than the diluent or intradermal with wheal ≥7 mm larger than the diluent control) within the last 4 years to fall pollen allergens present and prevalent in his/her geographic region.
* Signs and symptoms of nasal congestion (defined as stuffy or blocked nose) of at least mild severity (sign/symptom clearly present, but minimal awareness; easily tolerated) following the washout period (if applicable). Participant's diary evaluation must document at least mild symptoms for reflective and instantaneous scores on 4 consecutive days prior to randomization.
* Mean seated (after 5 minutes of rest) systolic/diastolic blood pressure ≤ 138/88 mmHg.
* Clinically acceptable physical exam and 12-lead ECG (recorded at 25 mm/s) that is clinically acceptable to the investigator.
* Free of any clinically significant disease that requires a physician's care and/or would interfere with trial evaluations, procedures, or participation.
* Agrees not to take monoamine oxidase inhibitors (MAOIs) from 14 days before trial participation until 14 days after the last dose of study drug.
* Capable of reading English.

Exclusion Criteria:

- Significant medical condition that is a contraindication to the use of phenylephrine, might

interfere with the trial, or requires treatment expected to affect blood pressure

* History or presence of hypertension
* Started allergen immunotherapy within 1 month of enrollment, will start immunotherapy during

the trial, or anticipates immunotherapy dose change during the trial

* Used Xolair (omalizumab) within 4 years prior to trial participation
* Known allergy or intolerance to phenylephrine, loratadine, or desloratadine
* History of rhinitis medicamentosa
* Documented evidence of acute or significant chronic sinusitis
* Clinically significant nasal disorders such as deviated septum and nasal polyposis
* Asthma, with the exception of mild intermittent asthma
* Have used systemic (oral, rectal, injectable), topical (up to 1% topical hydrocortisone

permitted), or nasal corticosteroids in the last 30 days

* Mentally or legally incapacitated, has significant emotional problems at the time of the Screening Visit or expected during the conduct of the study, or has a history of a clinically significant psychiatric disorder over the last 5 years. Those who have had situational depression may be enrolled in the study at the discretion of the investigator.
* History of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
* History of immunological disease or cancer within the past 5 years, with the exception of nonmelanoma skin cancer
* Positive drug screen (participants on prescribed medication resulting in a positive drug screen result may still be enrolled at the discretion of the investigator).
* Major surgery or participation in another investigational study within 30 days prior to the Screening Visit.
* Body mass index (BMI) ≥ 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 575 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

REFERENCES:
- [Derived] Meltzer EO, Ratner PH, McGraw T. Phenylephrine hydrochloride modified-release tablets for nasal congestion: a randomized, placebo-controlled trial in allergic rhinitis patients. Ann Allergy Asthma Immunol. 2016 Jan;116(1):66-71. doi: 10.1016/j.anai.2015.10.022. Epub 2015 Nov 7. PMID 26560899

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 29 centers in the United States;
  Study Period: August 2011 to October 2011
Groups:
- Phenylephrine: Phenylephrine hydrochloride, 30 mg extended-release tablets, one tablet every 12 hours for 7 days
- Placebo: Placebo to phenylephrine hydrochloride, 30-mg extended release tablets, one tablet every 12 hours for 7 days
Period: Overall Study
Arm/Group | Phenylephrine | Placebo
Started | 288 | 287
Completed | 288 | 286
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phenylephrine: Phenylephrine hydrochloride, 30-mg extended release tablets, one tablet every 12 hours for 7 days
- Total: Total of all reporting groups
Arm/Group | Phenylephrine | Placebo | Total
Number analyzed (Participants) | 288 | 287 | 575
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (11.64) | 40.1 (11.62) | 40.1 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 177 | 353
  Male | 112 | 110 | 222

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Daily Reflective Nasal Congestion Score
Description: The reflective assessment is a self-evaluation of the symptom severity over the preceding 12 hours. Baseline values were calculated as the mean from 4 consecutive 24-hour periods in which a symptom score was ≥1, prior to randomization. The nasal congestion score was calculated from data captured twice daily (morning and evening) in the participant's diary during the run-in and treatment periods. Participants rated congestion on a 4-point scale of severity: 0 = absent symptoms (no sign/symptom evident), 1 = mild symptoms (sign/symptom clearly present, but minimal awareness; easily tolerated), 2 = moderate symptoms (definite awareness of sign/symptom that is bothersome but tolerable), and 3 = severe symptoms (sign/symptom that is hard to tolerate; causes interference with activities of daily living and/or sleeping). The average of individual reflective nasal scores was reported as the daily reflective nasal congestion score over the entire treatment period.
Time Frame: Baseline and Days 1-7
Population: Efficacy analysis was performed on the intent-to-treat population (all randomized participants who received at least 1 dose of study medication). Number of participants evaluable in the placebo group at baseline was 287 and for the treatment period was 286.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Phenylephrine | Placebo
Number analyzed (Participants) | 288 | 287
Scores on a scale
  Baseline | 2.357 (0.5203) | 2.271 (0.5586)
  Change from Baseline for Entire Treatment Period | -0.394 (0.4880) | -0.412 (0.5383)

2. Secondary Outcome: Mean Change From Baseline in the Morning Reflective Symptom Assessment Score
Description: The reflective assessment is a self-evaluation of the symptom severity over the preceding 12 hours. Baseline values were calculated as the mean from 4 consecutive 24-hour periods in which a symptom score was ≥1, prior to randomization. The daily morning nasal congestion score was calculated from data captured daily (morning) in the participant's diary during the run-in and treatment periods. Participants rated congestion on a 4-point scale of severity: 0 = best and 3 = worst symptoms. The average of individual reflective nasal scores was reported as the daily reflective nasal congestion score over the entire treatment period.
Time Frame: Baseline and Days 1-7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Phenylephrine | Placebo
Number analyzed (Participants) | 288 | 287
Scores on a scale
  Baseline | 2.357 (0.5480) | 2.274 (0.5801)
  Entire Treatment Period | -0.403 (0.5420) | -0.425 (0.5868)

3. Secondary Outcome: Mean Change From Baseline in the Evening Reflective Symptom Assessment Score
Description: The reflective assessment is a self-evaluation of the symptom severity over the preceding 12 hours. Baseline values were calculated as the mean from 4 consecutive 24-hour periods in which a symptom score was ≥1, prior to randomization. The daily evening nasal congestion score was calculated from data captured daily (evening) in the participant's diary during the run-in and treatment periods. Participants rated congestion on a 4-point scale of severity: 0 = best and 3 = worst symptoms). The average of individual reflective nasal scores was reported as the daily reflective nasal congestion score over the entire treatment period.
Time Frame: Baseline and Days 1-7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Phenylephrine | Placebo
Number analyzed (Participants) | 288 | 287
Scores on a scale
  Baseline | 2.353 (0.5470) | 2.261 (0.5932)
  Entire Treatment Period | -0.403 (0.5424) | -0.424 (0.5894)

4. Secondary Outcome: Mean Change From Baseline in Daily Instantaneous Symptom Assessment Score
Description: The instantaneous assessment is a self-evaluation of the symptom severity at the moment of the assessment prior to the next dose. Baseline values were calculated as the mean from 4 consecutive 24-hour periods in which a symptom score was ≥1, prior to randomization. The daily nasal congestion score was calculated from data captured twice daily (morning and evening) in the participant's diary during the run-in and treatment periods. Participants rated congestion on a 4-point scale of severity: 0 = best and 3 = worst symptoms. The average of individual instantaneous nasal scores was reported as the daily instantaneous nasal congestion score over the entire treatment period.
Time Frame: Baseline and Days 1-7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Phenylephrine | Placebo
Number analyzed (Participants) | 288 | 286
Scores on a scale
  Baseline | 2.299 (0.5250) | 2.225 (0.5498)
  Entire Treatment Period | -0.311 (0.4663) | -0.366 (0.5265)

5. Secondary Outcome: Mean Change From Baseline in Daily Reflective Nasal Congestion Score Per Day
Description: The reflective assessment is a self-evaluation of the symptom severity over the preceding 12 hours. Baseline values were calculated as the mean from 4 consecutive 24-hour periods in which a symptom score was ≥1, prior to randomization. The nasal congestion score was calculated from data captured twice daily (morning and evening) in the participant's diary during the run-in and treatment periods. Participants rated congestion on a 4-point scale of severity: 0 = best and 3 = severe symptoms. The average of individual reflective nasal scores were reported as the daily reflective nasal congestion score for each day of the treatment period.
Time Frame: Baseline and Day 1, 2, 3, 4, 5, 6, and 7
Population: Efficacy analysis was performed on the intent-to-treat population (all randomized participants who received at least 1 dose of study medication). For the Phenylephrine Group, there were 287 evaluable participants on Day 1 and 288 on Days 2 - 7. For Placebo Group, there were 286 evaluable participants on Days 1, 2, 3, 4, 5, 6, and 285 on Day 7.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Phenylephrine | Placebo
Number analyzed (Participants) | 288 | 287
Scores on a scale
  Baseline | 2.357 (0.5203) | 2.271 (0.5586)
  Day 1 | -0.261 (0.5545) | -0.197 (0.6335)
  Day 2 | -0.302 (0.5248) | -0.321 (0.5721)
  Day 3 | -0.401 (0.6100) | -0.396 (0.6227)
  Day 4 | -0.395 (0.6234) | -0.492 (0.6942)
  Day 5 | -0.465 (0.6475) | -0.478 (0.6977)
  Day 6 | -0.461 (0.6918) | -0.488 (0.7444)
  Day 7 | -0.474 (0.7116) | -0.512 (0.7903)

6. Secondary Outcome: Mean Change From Baseline in Daily Instantaneous Symptom Assessment Score Per Day
Description: The instantaneous assessment is a self-evaluation of the symptom severity at the moment of the assessment prior to the next dose. Baseline values were calculated as the mean from 4 consecutive 24-hour periods in which a symptom score was ≥1, prior to randomization. The daily nasal congestion score was calculated from data captured twice daily (morning and evening) in the participant's diary during the run-in and treatment periods. Participants rated congestion on a 4-point scale of severity: 0 = best and 3 = worst symptoms. The average of individual instantaneous nasal scores was reported as the daily instantaneous nasal congestion score for each day of the treatment period.
Time Frame: Baseline and Day 1, 2, 3, 4, 5, 6, 7
Population: The Intent-To-Treat Population was used in this analysis. For the Phenylephrine Group, there were 287 evaluable participants on Day 1 and 288 on Day 2 - 7. For the Placebo Group, there were 286 evaluable participants on Days 1, 2, 3, 4, 5, 6 and 285 on Day 7.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Phenylephrine | Placebo
Number analyzed (Participants) | 288 | 287
Scores on a scale
  Baseline | 2.299 (0.5250) | 2.225 (0.5498)
  Day 1 | -0.192 (0.5809) | -0.200 (0.6451)
  Day 2 | -0.255 (0.5046) | -0.256 (0.5472)
  Day 3 | -0.307 (0.6206) | -0.373 (0.6548)
  Day 4 | -0.351 (0.6133) | -0.406 (0.6881)
  Day 5 | -0.359 (0.6432) | -0.406 (0.6632)
  Day 6 | -0.361 (0.6582) | -0.443 (0.7336)
  Day 7 | -0.352 (0.6698) | -0.476 (0.7829)

7. Secondary Outcome: Time to Maximal Phenylephrine Effect
Description: The time to maximal phenylephrine effect was defined as the earliest time that the nasal congestion symptom score in the Phenylephrine treatment group demonstrated the greatest numerical difference from the Placebo treatment group in change from baseline. The mean change from baseline scores for a Phenylephrine treatment arm and for the Placebo treatment arm at each timepoint of the treatment period (Day 1 morning, Day 1 evening, etc) was calculated. The difference between the Phenylephrine treatment arm and Placebo treatment arm mean at each timepoint of the treatment period was calculated. The time to maximal phenylephrine effect was the first timepoint at which the difference between the Phenylephrine treatment arm and the Placebo treatment arm was greatest. The results for the Placebo treatment arm are not presented as the result of this outcome measure is only relevant for the Phenylephrine treatment group.
Time Frame: Baseline up to Day 7
Population: All participants in the intent-to-treat population (all randomized participants who received at least 1 tablet of study medication).
Measure: Number; unit: Days
Groups:
- Phenylephrine: Phenylephrine hydrochloride 30 mg extended release tablets, one dose every 12 hours for 7 days
Arm/Group | Phenylephrine
Number analyzed (Participants) | 288
Days | 0.5

8. Secondary Outcome: Day 7 Mean Change From Baseline in Daily Instantaneous Symptom Assessment Score
Description: The instantaneous assessment is a self-evaluation of the symptom severity at the moment of the assessment prior to the next dose. Baseline values were calculated as the mean from 4 consecutive 24-hour periods in which a symptom score was ≥1, prior to randomization. The nasal congestion score was calculated from data captured twice daily (morning and evening) in the participant's diary during the run-in and treatment periods. Participants rated congestion on a 4-point scale of severity: 0 = best and 3 = worst symptoms). The average of individual instantaneous nasal scores was reported as the daily instantaneous nasal congestion score over the entire treatment period.
Time Frame: Baseline and Day 7
Population: Efficacy analysis was performed on the intent-to-treat population (all randomized participants who received at least 1 dose of study medication). Number of participants evaluable in the placebo group at baseline was 287 and at Day 7 was 285.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Phenylephrine | Placebo
Number analyzed (Participants) | 288 | 287
Scores on a scale
  Baseline | 2.299 (0.5250) | 2.225 (0.5498)
  Day 7 | -0.352 (0.6698) | -0.476 (0.7829)

9. Secondary Outcome: Mean Change From Baseline in Morning Predose Instantaneous Nasal Congestion Symptom Score
Description: The instantaneous assessment is a self-evaluation of the symptom severity at the moment of the assessment prior to the next dose. Baseline values were calculated as the mean from 4 consecutive 24-hour periods in which a symptom score was ≥1, prior to randomization. The nasal congestion score was calculated from data captured daily (morning) in the participant's diary during the run-in and treatment periods. Participants rated congestion on a 4-point scale of severity: 0 = best and 3 = worst symptoms. The average of individual morning instantaneous nasal scores was reported as the daily morning instantaneous nasal congestion score over the entire treatment period.
Time Frame: Baseline and Days 1-7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Phenylephrine | Placebo
Number analyzed (Participants) | 288 | 287
Scores on a scale
  Baseline | 2.313 (0.5518) | 2.264 (0.5816)
  Entire Treatment Period | -0.295 (0.5088) | -0.363 (0.5815)

10. Secondary Outcome: Mean Change From Baseline for the Morning Reflective Symptom Assessment Scores for Each Day During the Treatment Period.
Description: The reflective assessment is a self-evaluation of the symptom severity over the preceding 12 hours. Baseline values were calculated as the mean from 4 consecutive 24-hour periods in which a symptom score was ≥1, prior to randomization. The nasal congestion score was calculated from data captured daily (morning) in the participant's diary during the run-in and treatment periods. Participants rated congestion on a 4-point scale of severity: 0 = best and 3 = severe symptoms. The average of individual reflective nasal scores were reported as the daily reflective nasal congestion score for each day of the treatment period.
Time Frame: Baseline and Day 2, 3, 4, 5, 6, and 7
Population: The Intent-To-Treat Population was used in this analysis. For the Phenylephrine Group, there were 288 evaluable participants on Days 2 - 5 and 287 on Day 6. For the Placebo Group, there were 287 evaluable participants on Day 1, 286 on Days 2, 5, and 6 and 285 on Days 3, 4, and 7.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Phenylephrine | Placebo
Number analyzed (Participants) | 288 | 287
Scores on a scale
  Baseline | 2.357 (0.5480) | 2.274 (0.5801)
  Day 2 | -0.263 (0.5769) | -0.273 (0.6685)
  Day 3 | -0.402 (0.6723) | -0.380 (0.6932)
  Day 4 | -0.367 (0.7147) | -0.469 (0.7482)
  Day 5 | -0.451 (0.7214) | -0.480 (0.7631)
  Day 6 | -0.456 (0.7425) | -0.462 (0.8294)
  Day 7 | -0.478 (0.7830) | -0.489 (0.8515)

11. Secondary Outcome: Mean Change From Baseline for the Evening Reflective Symptom Assessment Scores for Each Day During the Treatment Period
Description: The reflective assessment is a self-evaluation of the symptom severity over the preceding 12 hours. Baseline values were calculated as the mean from 4 consecutive 24-hour periods in which a symptom score was ≥1, prior to randomization. The nasal congestion score was calculated from data captured daily (evening) in the participant's diary during the run-in and treatment periods. Participants rated congestion on a 4-point scale of severity: 0 = best and 3 = severe symptoms. The average of individual reflective nasal scores were reported as the daily reflective nasal congestion score for each day of the treatment period.
Time Frame: Baseline and Day 1, 2, 3, 4, 5, 6, and 7
Population: The Intent-To-Treat Population was used in this analysis. For the Phenylephrine Group, there were 288 evaluable participants on Day 5, 287 on Days 1, 3, 4, 6 and 286 on Day 2. For the Placebo Group, there were 287 evaluable participants on Day 1, 286 on Days 2, 5, 6, 285 on Days 3 and 7 and 284 on Day 4.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Phenylephrine | Placebo
Number analyzed (Participants) | 288 | 287
Scores on a scale
  Baseline | 2.353 (0.5470) | 2.261 (0.5932)
  Day 1 | -0.257 (0.5850) | -0.187 (0.6583)
  Day 2 | -0.343 (0.6732) | -0.362 (0.6729)
  Day 3 | -0.402 (0.7200) | -0.404 (0.7336)
  Day 4 | -0.420 (0.7294) | -0.511 (0.8180)
  Day 5 | -0.475 (0.7154) | -0.470 (0.7997)
  Day 6 | -0.463 (0.7593) | -0.509 (0.8143)
  Day 7 | -0.464 (0.7813) | -0.528 (0.8802)

12. Secondary Outcome: Mean Change From Baseline for the Morning Instantaneous Symptom Assessment Scores for Each Day During the Treatment Period
Description: The instantaneous assessment is a self-evaluation of the symptom severity at the moment of the assessment prior to the next dose. Baseline values were calculated as the mean from 4 consecutive 24-hour periods in which a symptom score was ≥1, prior to randomization. The daily nasal congestion score was calculated from data captured daily (morning) in the participant's diary during the run-in and treatment periods. Participants rated congestion on a 4-point scale of severity: 0 = best and 3 = worst symptoms. The average of individual instantaneous nasal scores was reported as the daily instantaneous nasal congestion score for each day of the treatment period.
Time Frame: Baseline and Day 2, 3, 4, 5, 6, and 7
Population: The Intent-To-Treat Population was used in this analysis. For the Phenylephrine Group, there were 288 evaluable participants on Days 1, 2, 3, 4, 5, 7 and 286 evaluable participants at Day 6. For the Placebo Group, there were 287 evaluable participants on Day 1, 286 on Days 3, 5, 6 and 285 on Days 2, 4, 7.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Phenylephrine | Placebo
Number analyzed (Participants) | 288 | 287
Scores on a scale
  Baseline | 2.313 (0.5518) | 2.264 (0.5816)
  Day 2 | -0.188 (0.5680) | -0.185 (0.6511)
  Day 3 | -0.285 (0.6888) | -0.373 (0.7389)
  Day 4 | -0.326 (0.7035) | -0.383 (0.7680)
  Day 5 | -0.326 (0.7201) | -0.387 (0.7617)
  Day 6 | -0.327 (0.7128) | -0.394 (0.8314)
  Day 7 | -0.319 (0.7488) | -0.462 (0.8618)

13. Secondary Outcome: Mean Change From Baseline for the Evening Instantaneous Symptom Assessment Scores for Each Day During the Treatment Period.
Description: The instantaneous assessment is a self-evaluation of the symptom severity at the moment of the assessment prior to the next dose. Baseline values were calculated as the mean from 4 consecutive 24-hour periods in which a symptom score was ≥1, prior to randomization. The daily nasal congestion score was calculated from data captured daily (evening) in the participant's diary during the run-in and treatment periods. Participants rated congestion on a 4-point scale of severity: 0 = best and 3 = worst symptoms. The average of individual instantaneous nasal scores was reported as the daily instantaneous nasal congestion score for each day of the treatment period.
Time Frame: Baseline and Day 1, 2, 3, 4, 5, 6, and 7
Population: Intent-To-Treat Population was used in this analysis. For the Phenylephrine Group, there were 288 evaluable participants on Days 5 and 7, 287 on Days 1, 3, 4 and 286 on Days 2 and 6. For the Placebo Group, there were 286 evaluable participants on Days 1, 2, 3, 5, 6 and 285 on Day 7 and 284 on Day 4.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Phenylephrine | Placebo
Number analyzed (Participants) | 288 | 287
Scores on a scale
  Baseline | 2.300 (0.5612) | 2.189 (0.5878)
  Day 1 | -0.193 (0.5888) | -0.164 (0.6415)
  Day 2 | -0.344 (0.6768) | -0.332 (0.7020)
  Day 3 | -0.349 (0.7591) | -0.378 (0.7773)
  Day 4 | -0.395 (0.7529) | -0.434 (0.8079)
  Day 5 | -0.408 (0.7558) | -0.430 (0.7714)
  Day 6 | -0.424 (0.7584) | -0.497 (0.8122)
  Day 7 | -0.401 (0.7865) | -0.495 (0.8645)

14. Secondary Outcome: Rhinoconjunctivitis Quality of Life Questionnaire With Standardized Activities (RQLQ)
Description: The RQLQ is a disease-specific quality of life questionnaire developed to measure the physical, emotional, and social problems in adults with rhinoconjunctivitis. Questions were divided into 7 domains: sleep (3 questions), non-hay fever symptoms (7 questions), practical problems (3
  questions), nasal symptoms (4 questions), eye symptoms (4 questions), and activities (3 questions), and emotions (4 questions). Individual items within the RQLQ are equally weighted. The questionnaire is analyzed directly from the scores recorded and the results are expressed as the mean score for each of the domains (i.e., domain scores range from 0 to 6). Six represents the greatest impairment and 0 represents the least impairment. Overall quality of life score is the mean score for all domains.
Time Frame: Up to Day 8
Population: The Intent-To-Treat Population was used in this analysis. There were 285 evaluable participants for the Placebo Group at Day 8.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Phenylephrine | Placebo
Number analyzed (Participants) | 288 | 287
Scores on a scale
  Baseline | 3.6 (1.28) | 3.5 (1.28)
  Day 8 | -0.8 (1.15) | -0.9 (1.13)

ADVERSE EVENTS:
Time Frame: Up to Day 31
Description: Safety analyses was performed on the Safety Population, which was defined as all
  randomized subjects who received at least 1 dose of study medication.
Arm/Group | Phenylephrine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/288 | 0/287
Other Adverse Events (participants affected / at risk) | 0/288 | 0/287

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts,

manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.